CLINICAL TRIAL: NCT02335411
Title: A Phase II Clinical Trial of Pembrolizumab as Monotherapy and in Combination With Cisplatin+5-Fluorouracil in Subjects With Recurrent or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (KEYNOTE-059)
Brief Title: A Study of Pembrolizumab (MK-3475) in Participants With Recurrent or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (MK-3475-059/KEYNOTE-059)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-059; MK-3475-059 (Other: Merck); KEYNOTE-059 (Other: Merck); 2014-003574-16 (EudraCT Number)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric cancer; Gastroesophageal junction cancer; Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Pembrolizumab monotherapy, previously treated (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W)
  Interventions: Biological: pembrolizumab
- Cohort 2: Pembrolizumab combination therapy, treatment naive (Experimental): Participants receive pembrolizumab 200 mg IV each 3-week cycle (Q3W) + cisplatin 80 mg/m^2 IV Q3W for up to 6 cycles + 5-FU 800 mg/m^2 IV on Days 1-5 every 3 weeks or (Japan only) capecitabine 1000 mg/m^2 orally, twice per day (BID) on Days 1-14 of each 3-week cycle
  Interventions: Biological: pembrolizumab; Drug: cisplatin; Drug: 5-FU; Drug: capecitabine
- Cohort 3: Pembrolizumab monotherapy, treatment naive, PD-L1 positive (Experimental): Programmed death-ligand 1 (PD-L1) positive participants receive pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W)
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475
Drug: cisplatin — IV infusion
  Other Names: PLATINOL®
  Arms: Cohort 2: Pembrolizumab combination therapy, treatment naive
Drug: 5-FU — IV infusion
  Other Names: ADRUCIL®
  Arms: Cohort 2: Pembrolizumab combination therapy, treatment naive
Drug: capecitabine — oral tablets
  Other Names: XELODA®
  Arms: Cohort 2: Pembrolizumab combination therapy, treatment naive

SUMMARY:
This is a study of pembrolizumab (MK-3475) for advanced gastric or gastroesophageal junction adenocarcinoma; pembrolizumab will be given as monotherapy to participants who have had previous treatment or who are treatment-naïve; pembrolizumab will also be evaluated as combination therapy with cisplatin and 5-Fluorouracil (5-FU) or (Japan only) capecitabine in treatment-naïve participants. The primary study hypothesis is that pembrolizumab will provide a clinically meaningful Overall Response Rate (ORR).

DETAILED DESCRIPTION:
This study will have 3 cohorts. In Cohort 1, participants who have received at least two prior therapies for their advanced disease will receive monotherapy with pembrolizumab. In Cohort 2, participants who have not received any previous therapy for their disease will receive pembrolizumab in combination with cisplatin and 5-FU or (Japan only) capecitabine. In Cohort 3, participants who have not received any previous therapy and who have programmed death ligand 1 (PD-L1)-positive tumors will receive pembrolizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria - Cohort 1:

* Received and progressed on ≥2 prior chemotherapy regimens for their advanced disease; prior regimen must have included a cisplatin and a fluoropyridine
* Human epidermal growth factor receptor 2 (HER-2/neu) negative, or, if HER2/neu positive, must have previously received treatment with trastuzumab

Inclusion Criteria - Cohort 2 or 3:

* HER2/neu negative
* Has not received prior systemic anti-cancer therapy for their advanced carcinoma (systemic therapy received in the neoadjuvant and adjuvant setting does not count)

Inclusion Criteria - All Participants:

* Histologically- or cytologically-confirmed recurrent or metastatic gastric or gastroesophageal junction adenocarcinoma that is considered incurable by local therapies
* Willing to provide tissue for PD-L1 biomarker analysis from newly-obtained and/or archival tissue
* Measurable disease based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 3 days prior to first dose of study drug
* Life expectancy of at least 3 months
* Female participants of childbearing potential should have a negative pregnancy test and be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study drug (180 days for participants receiving cisplatin + 5FU)
* Male participants should agree to use an adequate method of contraception starting with the first dose through 120 days after the last dose of study drug (180 days for participants receiving cisplatin + 5FU)
* Adequate organ function

Exclusion Criteria - All Participants:

* Currently participating and receiving study therapy or participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of study drug
* Active autoimmune disease that has required systemic treatment in past 2 years
* Immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Weight loss >10% over 2 months prior to first dose of study drug
* Clinical evidence of ascites by physical exam
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or not recovered from AEs due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered from AEs due to a previously administered agent
* Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Known history of, or any evidence of active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug (180 days for participants receiving cisplatin + 5FU)
* Prior therapy with an anti-programmed death-1 (PD-1), anti-PD-L1, or anti-PD-L2 agent
* Human immunodeficiency virus (HIV)
* Hepatitis B or C
* Received live vaccine within 30 days of planned start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Janjigian YY, Cecchini M, Shitara K, Enzinger PC, Wainberg ZA, Chau I, Satoh T, Lee J, Nebozhyn M, Loboda A, Kobie J, Vajdi A, Shih CS, Cristescu R, Cao ZA. Genomic Landscape of Late-Stage Gastric Cancer: Analysis From KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Studies. JCO Precis Oncol. 2025 Mar;9:e2400456. doi: 10.1200/PO-24-00456. Epub 2025 Mar 21. PMID 40117530
- [Derived] Topp BG, Channavazzala M, Mayawala K, De Alwis DP, Rubin E, Snyder A, Wolchok JD, Ribas A. Tumor dynamics in patients with solid tumors treated with pembrolizumab beyond disease progression. Cancer Cell. 2023 Sep 11;41(9):1680-1688.e2. doi: 10.1016/j.ccell.2023.08.004. PMID 37699333
- [Derived] Muro K, Shitara K, Yamaguchi K, Yoshikawa T, Satake H, Hara H, Sugimoto N, Machida N, Goto M, Kawakami H, Amagai K, Omuro Y, Esaki T, Hironaka S, Nishina T, Komatsu Y, Matsubara H, Shiratori S, Han S, Satoh T, Ohtsu A. Efficacy of Pembrolizumab Monotherapy in Japanese Patients with Advanced Gastric or Gastroesophageal Junction Cancer. J Gastrointest Cancer. 2023 Sep;54(3):951-961. doi: 10.1007/s12029-023-00920-9. Epub 2023 Apr 10. PMID 37037952
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Chao J, Fuchs CS, Shitara K, Tabernero J, Muro K, Van Cutsem E, Bang YJ, De Vita F, Landers G, Yen CJ, Chau I, Elme A, Lee J, Ozguroglu M, Catenacci D, Yoon HH, Chen E, Adelberg D, Shih CS, Shah S, Bhagia P, Wainberg ZA. Assessment of Pembrolizumab Therapy for the Treatment of Microsatellite Instability-High Gastric or Gastroesophageal Junction Cancer Among Patients in the KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Clinical Trials. JAMA Oncol. 2021 Jun 1;7(6):895-902. doi: 10.1001/jamaoncol.2021.0275. PMID 33792646
- [Derived] Bang YJ, Kang YK, Catenacci DV, Muro K, Fuchs CS, Geva R, Hara H, Golan T, Garrido M, Jalal SI, Borg C, Doi T, Yoon HH, Savage MJ, Wang J, Dalal RP, Shah S, Wainberg ZA, Chung HC. Pembrolizumab alone or in combination with chemotherapy as first-line therapy for patients with advanced gastric or gastroesophageal junction adenocarcinoma: results from the phase II nonrandomized KEYNOTE-059 study. Gastric Cancer. 2019 Jul;22(4):828-837. doi: 10.1007/s10120-018-00909-5. Epub 2019 Mar 25. PMID 30911859
- [Derived] Fuchs CS, Doi T, Jang RW, Muro K, Satoh T, Machado M, Sun W, Jalal SI, Shah MA, Metges JP, Garrido M, Golan T, Mandala M, Wainberg ZA, Catenacci DV, Ohtsu A, Shitara K, Geva R, Bleeker J, Ko AH, Ku G, Philip P, Enzinger PC, Bang YJ, Levitan D, Wang J, Rosales M, Dalal RP, Yoon HH. Safety and Efficacy of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Clinical KEYNOTE-059 Trial. JAMA Oncol. 2018 May 10;4(5):e180013. doi: 10.1001/jamaoncol.2018.0013. Epub 2018 May 10. PMID 29543932
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants of at least 18 years of age with recurrent or metastatic gastric or gastro-esophageal junction (GEJ) adenocarcinoma were enrolled in this study.
Pre-assignment Details: 318 participants were originally allocated to the study. No study information was collected from 3 participants, who were excluded from all analyses, including disposition.
  Per protocol, response/progression or adverse events during the second pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures respectively.
Groups:
- Cohort 1: Pembrolizumab Monotherapy, Previously Treated: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for up to 52 months. Eligible participants allocated to the pembrolizumab first course, who stopped pembrolizumab with stable disease (SD) or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg of each 3 week cycle for up to 17 cycles up to approximately an additional year.
- Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive: Participants received pembrolizumab 200 mg IV each 3-week cycle (Q3W) for up to 40 months + cisplatin 80 mg/m^2 IV Q3W for up to 6 cycles + 5-Fluorouracil (5-FU) 800 mg/m^2 IV on Days 1-5 every 3 weeks or (Japan only) capecitabine 1000 mg/m^2 orally, twice per day (BID) on Days 1-14 of each 3-week cycle. Eligible participants allocated to the pembrolizumab first course, who stopped pembrolizumab with SD or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg of each 3 week cycle for up to 17 cycles up to approximately an additional year.
- Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive: Programmed death-ligand 1 (PD-L1) positive participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 52 months. Eligible participants allocated to the pembrolizumab first course, who stopped pembrolizumab with SD or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg of each 3 week cycle for up to 17 cycles up to approximately an additional year.
Period: Overall Study
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Started (First Course Pembrolizumab) | 259 | 25 | 31
Second Course Pembrolizumab | 3 | 1 | 2
Completed | 0 | 0 | 0
Not Completed | 259 | 25 | 31
Not completed — Death | 223 | 22 | 26
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 3
Not completed — Sponsor Decision | 12 | 3 | 2
Not completed — Adverse Event | 9 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive | Total
Number analyzed (Participants) | 259 | 25 | 31 | 315
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (11.4) | 58.8 (16.6) | 60.3 (11.2) | 60.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 9 | 12 | 82
  Male | 198 | 16 | 19 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 1 | 3 | 21
  Not Hispanic or Latino | 228 | 23 | 28 | 279
  Unknown or Not Reported | 14 | 1 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 41 | 17 | 15 | 73
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 0 | 5
  White | 200 | 8 | 16 | 224
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 11 | 0 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with the study drug. The number of participants who experienced at least one AE is presented. Per protocol, the number of participants who experienced at least one AE during first course pembrolizumab treatment is presented.
Time Frame: Up to approximately 65 months
Population: All enrolled participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 259 | 25 | 31
Participants | 248 | 25 | 31

2. Primary Outcome: Number of Participants Discontinuing Study Drug Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with the study drug. The number of participants who discontinued study drug due to an AE is presented. Per protocol, the number of participants who discontinued drug during first course pembrolizumab treatment is presented.
Time Frame: Up to approximately 52 months
Population: All enrolled participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 259 | 25 | 31
Participants | 18 | 4 | 0

3. Primary Outcome: Objective Response Rate (ORR) For All Participants in Cohorts 1 and 3
Description: The Objective Response Rate (ORR) was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by central radiology review. The percentage of all participants (regardless of programmed death-ligand 1 [PD-L1] tumor status) in Cohorts 1 and 3 who had a CR or PR during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants in Cohorts 1 and 3 who received ≥1 dose of study drug. Per protocol, Cohort 2 was not included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 259 | 0 | 31
Percentage of Participants | 11.6 [8.0 to 16.1] |  | 22.6 [9.6 to 41.1]

4. Primary Outcome: Objective Response Rate For PD-L1 Positive Participants in Cohorts 1 and 3
Description: The ORR was defined as the percentage of participants in the analysis population who had a CR or PR (CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, as assessed by central radiology review. The percentage of all participants in Cohorts 1 and 3 with PD-L1+ tumor status who experienced a CR or PR during first course pembrolizumab treatment per protocol, is presented. Note: All participants in Cohort 3 had a PD-L1-positive tumor status.
Time Frame: Up to approximately 75 months
Population: All enrolled participants in Cohorts 1 and 3 with a positive PD-L1 tumor status who received ≥1 dose of study drug. Per protocol, Cohort 2 was not included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 148 | 0 | 31
Percentage of Participants | 15.5 [10.1 to 22.4] |  | 22.6 [9.6 to 41.1]

5. Secondary Outcome: Objective Response Rate (ORR) For All Participants in Cohort 2
Description: The Objective Response Rate (ORR) was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by central radiology review. The percentage of all participants (regardless of PD-L1 tumor status) in Cohort 2 who had a CR or PR during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants in Cohort 2 who received ≥1 dose of study drug. Per protocol, Cohorts 1 and 3 were not included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 0 | 25 | 0
Percentage of Participants |  | 60.0 [38.7 to 78.9] |

6. Secondary Outcome: Objective Response Rate For PD-L1 Positive Participants in Cohort 2
Description: The ORR was defined as the percentage of participants in the analysis population who had a CR or PR (CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, as assessed by central radiology review. The percentage of participants in Cohort 2 with PD-L1+ tumor status who experienced a CR or PR during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants in Cohort 2 with a positive PD-L1 tumor status who received ≥1 dose of study drug. Per protocol, Cohorts 1 and 3 were not included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 0 | 15 | 0
Percentage of Participants |  | 73.3 [44.9 to 92.2] |

7. Secondary Outcome: Duration of Response (DOR) For All Participants
Description: Duration of Response (DOR) was defined as the time from first documented evidence of CR or PR (CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, based on central imaging vendor assessment, until disease progression (PD) or death, whichever occurred first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Participants who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment. The DOR for all participants (regardless of PD-L1 tumor status) during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants who received ≥1 dose of study drug and demonstrated a confirmed response (CR or PR).
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 30 | 15 | 7
Months | 16.1 [2.4 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 4.6 [2.6 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 38.0 [2.1 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

8. Secondary Outcome: Duration of Response For PD-L1 Positive Participants
Description: DOR was defined as the time from first documented evidence of CR or PR (CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, based on central imaging vendor assessment, until disease progression (PD) or death, whichever occurred first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Participants who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment. The DOR for only PD-L1 positive participants during first course pembrolizumab treatment per protocol, is presented. Note: All participants in Cohort 3 had a PD-L1-positive tumor status.
Time Frame: Up to approximately 75 months
Population: All enrolled participants with a positive PD-L1 tumor status who received ≥1 dose of study drug and demonstrated a confirmed response (CR or PR).
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 23 | 11 | 7
Months | NA [NA to NA] — NA = median, upper and lower limits not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 4.6 [3.2 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 38.0 [2.1 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

9. Secondary Outcome: Progression-Free Survival (PFS) For All Participants
Description: Progression-Free Survival (PFS) was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. The PFS for all participants (regardless of PD-L1 tumor status) during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 259 | 25 | 31
Months | 2.0 [2.0 to 2.0] | 6.6 [5.9 to 10.6] | 2.9 [2.0 to 6.0]

10. Secondary Outcome: Progression-Free Survival For PD-L1 Positive Participants
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. The PFS for only PD-L1 positive participants during first course pembrolizumab treatment per protocol, is presented. Note: All participants in Cohort 3 had a PD-L1-positive tumor status.
Time Frame: Up to approximately 75 months
Population: All enrolled participants with a positive PD-L1 tumor status who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 148 | 15 | 31
Months | 2.1 [2.0 to 2.1] | 6.5 [4.7 to 7.9] | 2.9 [2.0 to 6.0]

11. Secondary Outcome: Overall Survival (OS) For All Participants
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. The OS for all participants (regardless of PD-L1 tumor status) during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 259 | 25 | 31
Months | 5.5 [4.2 to 6.7] | 13.8 [8.6 to 25.6] | 20.7 [10.0 to 29.8]

12. Secondary Outcome: Overall Survival For PD-L1 Positive Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. The OS for only PD-L1 positive participants during first course pembrolizumab treatment per protocol, is presented. Note: All participants in Cohort 3 had a PD-L1-positive tumor status.
Time Frame: Up to approximately 75 months
Population: All enrolled participants with a positive PD-L1 tumor status who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 148 | 15 | 31
Months | 5.8 [4.4 to 7.8] | 11.1 [5.4 to 22.3] | 20.7 [10.0 to 29.8]

13. Secondary Outcome: Disease Control Rate (DCR) For All Participants
Description: Disease Control Rate (DCR) was defined as the percentage of participants in the analysis population who had a CR or a PR (CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions) or stable disease (SD); (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) for ≥6 months, (for Cohort 1 ≥2 months) as assessed by central radiology review. The percentage of all participants (regardless of PD-L1 tumor status) who had a CR or PR or SD during first course pembrolizumab treatment per protocol, is presented.
Time Frame: Up to approximately 75 months
Population: All enrolled participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 259 | 25 | 31
Percentage of Participants | 27.0 [21.7 to 32.9] | 80.0 [59.3 to 93.2] | 32.3 [16.7 to 51.4]

14. Secondary Outcome: Disease Control Rate For PD-L1 Positive Participants
Description: DCR was defined as the percentage of participants in the analysis population who had a CR or a PR (CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions) or stable disease (SD); (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) for ≥6 months, (for Cohort 1 ≥2 months) as assessed by central radiology review. The percentage of participants with PD-L1+ tumor status who experienced a CR or PR or SD during first course pembrolizumab treatment per protocol, is presented. Note: All participants in Cohort 3 had a PD-L1-positive tumor status.
Time Frame: Up to approximately 75 months
Population: All enrolled participants with a positive PD-L1 tumor status who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Pembrolizumab Monotherapy, Previously Treated | Cohort 2: Pembrolizumab Combination Therapy, Treatment Naive | Cohort 3: Pembrolizumab Monotherapy, Treatment Naive, PD-L1 Positive
Number analyzed (Participants) | 148 | 15 | 31
Percentage of Participants | 33.1 [25.6 to 41.3] | 80.0 [51.9 to 95.7] | 32.3 [16.7 to 51.4]

ADVERSE EVENTS:
Time Frame: Up to approximately 75 months
Description: The population analyzed for all-cause mortality consisted of all allocated participants. The population for AEs consisted of all allocated participants who received ≥1 dose of study drug. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Therefore the following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression.
Groups:
- Cohort 1 First Course: Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 52 months.
- Cohort 2 First Course: Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 40 months + cisplatin 80 mg/m^2 IV Q3W for up to 6 cycles + 5-FU 800 mg/m^2 IV on Days 1-5 every 3 weeks or (Japan only) capecitabine 1000 mg/m^2 orally, BID on Days 1-14 of each 3-week cycle.
- Cohort 3 First Course: PD-L1 positive participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 52 months
- Cohort 1 Second Course: Eligible participants allocated to the pembrolizumab first course in Cohort 1 who stopped pembrolizumab with stable disease (SD) or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg on Day 1 of each 3 week cycle (Q3W) for up to 17 cycles up to approximately an additional year.
- Cohort 2 Second Course: Eligible participants allocated to the pembrolizumab first course in Cohort 2 who stopped pembrolizumab with SD or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg on Day 1 of each 3 week cycle (Q3W) for up to 17 cycles up to approximately an additional year.
- Cohort 3 Second Course: Eligible participants allocated to the pembrolizumab first course in Cohort 3 who stopped pembrolizumab with SD or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg on Day 1 of each 3 week cycle (Q3W) for up to 17 cycles up to approximately an additional year.
Arm/Group | Cohort 1 First Course | Cohort 2 First Course | Cohort 3 First Course | Cohort 1 Second Course | Cohort 2 Second Course | Cohort 3 Second Course
All-Cause Mortality (participants affected / at risk) | 244/259 | 21/25 | 26/31 | 1/3 | 1/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 119/259 | 11/25 | 15/31 | 0/3 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 237/259 | 25/25 | 31/31 | 0/3 | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 First Course (N=259) | Cohort 2 First Course (N=25) | Cohort 3 First Course (N=31) | Cohort 1 Second Course (N=3) | Cohort 2 Second Course (N=1) | Cohort 3 Second Course (N=2)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse uveal melanocytic proliferation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal intramural haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (6) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 First Course (N=259) | Cohort 2 First Course (N=25) | Cohort 3 First Course (N=31) | Cohort 1 Second Course (N=3) | Cohort 2 Second Course (N=1) | Cohort 3 Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 58 (69) | 11 (13) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (7) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 9 (12) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (10) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 10 (10) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 24 (24) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 15 (15) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 49 (56) | 3 (3) | 8 (13) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 19 (25) | 4 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 16 (18) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 52 (57) | 14 (22) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 46 (55) | 14 (18) | 8 (13) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 31 (36) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (12) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 65 (74) | 15 (22) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 10 (10) | 17 (29) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 36 (44) | 10 (23) | 6 (12) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 24 (26) | 4 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 93 (105) | 10 (13) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 4 (5) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 7 (7) | 5 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 9 (9) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 43 (57) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 25 (35) | 6 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (10) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 14 (19) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 30 (34) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 31 (32) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 13 (15) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 13 (30) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 38 (41) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 3 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 73 (81) | 13 (22) | 11 (14) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 15 (20) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (29) | 3 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 24 (24) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (13) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 23 (26) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (14) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (58) | 3 (3) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (38) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (12) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 17 (17) | 4 (5) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 6 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (13) | 5 (5) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 15 (18) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 17 (20) | 9 (9) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (50) | 2 (2) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (43) | 1 (2) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (18) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 33 (39) | 4 (7) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 31 (33) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 14 (20) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 10 (12) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT02335411/Prot_SAP_000.pdf